CLINICAL TRIAL: NCT01292382
Title: Effects of rTMS on the Cognition of Elderly With Cognitive Impairment no Dementia ( CIND )
Brief Title: Effects of rTMS on the Cognition of Elderly With Mild Memory Complaints
Acronym: TMSMemOld
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: University of Sao Paulo General Hospital, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rTMSCogOld
Record Dates: First submitted 2010-10-05; First posted 2011-02-09 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2010-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Elderly; Memory; Cognition; Repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS versus Sham (Sham Comparator): rTMS: active coil Sham: inactive coil
  Interventions: Device: Repetitive transcranial magnetic stimulation
- rTMS versus sham (Active Comparator): rTMS group: active coil Sham group: inactive coil
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Intensity: 110% of motor threshold Frequency: 10 Hz Number of trains: 40 trains Duration of trains: 5 seconds Interval: 25 seconds Number of sessions: 10 sessions Duration of intervention: two consecutive weeks
  Other Names: Active rTMS group; Sham rTMS group
Device: Repetitive transcranial magnetic stimulation — Intensity: 110% of motor threshold Frequency: 10 Hz Number of trains: 40 Duration of trains: 5 seconds Interval inter trains: 25 seconds Number of pulses each session: 2.000 Total number of pulses: 20.000
  Other Names: Arm 1: Active rTMS; Arm 2: Sham rTMS

SUMMARY:
Memory is constituted by a set of mental abilities of information processing that will be available at a later time. Flawless performance depends on several brain systems and other cognitive domains. Normal aging is characterized by cognitive deficits that may worsen the production capacity and quality of life. Such deficits represent variations of normal , and may stabilize,or even better progress. Include multiple cognitive domains, such as working and episodic memory, and attention. Despite the heterogeneity of the nature and severity of these deficits, common characteristics were observed in neuropsychological assessment of that population, for example, reduction in processing speed. There is an important gap in the therapeutic approach of these individuals.

Transcranial magnetic stimulation (TMS) is a noninvasive and promising intervention, with potential to improve memory and cognition activating networks that operate on memory or other networks that interfere with cognitive performance. The technique relies on generating a variable magnetic field originated from an alternating electric current applied to the human skull reaching focal cortical regions.

This study is a sham-controlled clinical trial, randomized, double-blind study. It will be evaluated the effects of repetitive transcranial magnetic stimulation (rTMS) on global cognition (memory, attention, language, executive functions, planning, logical reasoning, calculation and visual-spatial perception), especially memory, of elderly individuals with mild cognitive impairment, included in the domain of cognitive impairment no dementia (CIND).

DETAILED DESCRIPTION:
Subjects:

I. Eligibility criteria:

1. Male and female participants
2. Older adults aged 60-74 years
3. Education ≥ 4 years
4. Performance on neuropsychological tests below normal for age and education
5. Availability to attend the sessions of the application of TMS and neuropsychological assessments
6. Signing an informed consent by the participant or his guardian

II. No eligibility criteria:

1. Prior diagnosis of dementia
2. Any psychiatric disorder, except for mild depression in remission for at least 6 months. Shall be excluded those with scores > 12 on the Hamilton Depression Scale
3. History of neurosurgery and implantation of metal clips, head trauma, implantation of cardiac pacemakers, stroke, transient ischemic attack, cardiac surgery
4. Clinical or neurological diseases with impact on cognitive ability
5. Neurodegenerative central nervous system disease(eg. Parkinson Disease)
6. Alcohol and other drug abstinence for less than one year
7. Use of psychotropic medications (anticholinergic, mood stabilizers, neuroleptics), except for antidepressants
8. Chronic use of benzodiazepines with abstinence for less than 6 months
9. Severe uncontrolled organic disease that might interfere with the conduct of the study, such as cancer, congestive heart disease, digestive disorders, diabetes mellitus type I or type II, dyslipidemia etc.
10. Sensory impairments(to guarantee a adequate performance in the tests to evaluate cognitive functions)
11. Magnetic resonance imaging of the brain with evidence of lacunar or large vessels infarctions, cerebral hemorrhage

13. Hachinski Ischemic score of > 7 (or modified by Loeb > 5) 14. Any other condition that in the opinion of the investigator becomes problematic inclusion of the patient in a trial of this nature, as well as patients who do not adhere or do not cooperate.

III. Outcome measures:

Will be considered as an outcome measure a variation greater than or equal to 10% compared to baseline scores of neuropsychological tests, which will be applied on three occasions: immediately before (T0), after treatment (T2) and 4 weeks after the end of it (T3).

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes
* Aged between 60 and 74 years
* Schooling ≥ 4 years
* Performance on neuropsychological tests of up to 1.5 standard deviations below normal for age and education
* Signing an informed consent by the participant or his guardian.

Exclusion Criteria:

* Prior diagnosis of dementia.
* Any psychiatric disorder, except for mild depression for at least six months.
* Shall be excluded those with scores> 12 on the Hamilton scale.
* History of neurosurgery and implantation of metal clips, head trauma, implantation of cardiac pacemakers, stroke, transient ischemic attack, cardiac surgery
* Clinical or neurological diseases with an impact on cognitive ability
* Neurodegenerative central nervous system (eg Parkinson's disease)
* Alcohol and other drug dependency with abstinence for less than a year
* Use of psychotropic medications (anticholinergic, mood stabilizers, neuroleptics), except for antidepressants
* Chronic use of benzodiazepines with abstinence for less than six months
* Use of vitamin supplements (multivitamins, folic acid, vitamin B12), ginkgo biloba
* Severe uncontrolled organic disease that could interfere in the conduct of the study, such as cancer, heart disease, digestive disorders, diabetes mellitus type I or type II, uncontrolled dyslipidemia etc.
* Sensory disabilities, intellectual, preventing them from adequately perform the necessary tests to assess cognitive function
* Cerebrovascular disease based on Hachinsky score.
* History of head trauma.
* Any other condition that in the opinion of the investigator makes problematic the inclusion of the patient in a trial of this nature, as well as patients who do not adhere or not to cooperate.
* Worsening of the primary symptoms during the treatment.

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Repetitive transcranial magnetic stimulation improves memory in elderly with memory complaints | Neuropsychological tests: T1 - effects after rTMS, and T2: 4 weeks after rTMS
  Neuropsychological tests - RBMT (Rivermead Behavioral and Memory Test)

SECONDARY OUTCOMES:
Repetitive transcranial magnetic stimulation improves global cognition of elderly with memory complaints | Neuropsychological tests: T1 - effects after rTMS, and T2: 4 weeks after rTMS
  Performance on neuropsychological tests - STROOP, Trails 1 and 2, mini mental status exam (MMSE), clock drawing test, Wechsler, WAISS III, verbal fluency.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Marcolin, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil